CLINICAL TRIAL: NCT06974552
Title: The Effect of Different Support Surface Applications on Pressure Injury and Pain in Patients Undergoing Robotic Surgery
Brief Title: The Effect of Different Support Surface Applications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ukke Karabacak, Principal investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATADEK-2025/06
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pressure Incidence Prevention; Pain
Keywords: pressure injury; robotic surgery; deep trendelenburg position; pain
MeSH Terms: conditions — Pain; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Microbead-Filled Support Surface) (Experimental): Patients undergoing robotic surgery in the deep Trendelenburg position who received microbead-filled support surfaces applied to the shoulder areas.
  Interventions: Procedure: microbead-filled support surfaces
- Control Group (gel support surfaces ) (Other): Patients undergoing robotic surgery in the deep Trendelenburg position who received gel support surfaces applied to the shoulder areas.
  Interventions: Procedure: Jel support surfaces

INTERVENTIONS:
Procedure: microbead-filled support surfaces — Patients will undergo a preoperative pressure injury risk assessment. After the induction of general anesthesia, a multilayer silicone wound dressing will be applied to the shoulder area. The shoulder will then be supported using microbead-filled support surfaces. This support surface will remain in place throughout the duration of the surgery.
  Arms: Experimental Group (Microbead-Filled Support Surface)
Procedure: Jel support surfaces — Patients will undergo a preoperative pressure injury risk assessment. After the induction of general anesthesia, a multilayer silicone wound dressing will be applied to the shoulder area. The shoulder will then be supported using jel support surfaces. This support surface will remain in place throughout the duration of the surgery.
  Arms: Control Group (gel support surfaces )

SUMMARY:
This study was designed as a randomized controlled experimental study to compare the effects of two support surfaces-gel pads (used in routine practice) and microbead-filled pads-placed under the shoulders in the steep Trendelenburg position during robotic surgery, on the development of pressure injuries and pain.

DETAILED DESCRIPTION:
Safe and procedure-specific patient positioning is a critical component of successful surgical outcomes. In robotic surgeries, particularly those involving the lower pelvic region, the steep Trendelenburg position is frequently used to optimize surgical exposure. However, as the angle of the Trendelenburg position increases and the patient remains in this posture for a prolonged period, the risk of adverse events such as nerve injuries, pressure injuries, and deep tissue ischemia also increases.

Unlike traditional surgeries where repositioning the patient may be possible during the procedure, robotic surgeries do not allow for intraoperative repositioning due to the fixed docking of robotic arms. Consequently, safe and effective positioning strategies are essential to prevent patient movement and minimize the risk of skin and soft tissue damage.

The current systems used for managing patients in the steep Trendelenburg position are suboptimal. There is limited evidence in the literature regarding the incidence and prevention of pressure injuries associated with this specific position during robotic surgery. Prolonged immobility in this posture increases friction and pressure at contact surfaces, which can lead to pressure-related injuries.

The use of appropriate support surfaces is therefore vital to reduce the risk of such injuries. This study aims to address this gap by evaluating and comparing different support surfaces placed under the shoulders during robotic surgery in the steep Trendelenburg position, with a focus on their effects on pressure injury development and postoperative pain.

Hypotheses of the study H1: The use of microbead-filled support surfaces under the shoulders is superior to gel support surfaces in preventing pressure injuries and pain.

H2: The use of gel support surfaces under the shoulders is superior to microbead-filled support surfaces in preventing pressure injuries and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo robotic surgery in the lower pelvic region in the steep Trendelenburg position
* Patients aged 18 years and older

Exclusion Criteria:

* Patients with existing pressure injuries
* Patients with communication barriers
* Patients with skin anomalies that interfere with skin assessment
* Patients requiring conversion to open surgery during the procedure
* Patients whose position is changed during surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in the pressure injury condition | At the time of admission to the operating room, immediately after surgery, one hour after surgery, 12 hour after surgery, 24 hour after surgery. The change in this time intervals will be assessed.
  The presence or absence of pressure injuries in patients will be assessed. If a pressure injury is present, it will be staged accordingly. Pressure injury assessment will be conducted in accordance with the guidelines of the European Pressure Ulcer Advisory Panel (EPUAP) and the National Pressure Ulcer Advisory Panel (NPUAP)
Change in the pain level | Pain will be assessed every 15 minutes during the first two hours after surgery, and then every 30 minutes for the following one hour.The change in this time intervals will be assessed.
  The patient's pain will be assessed using the Visual Analog Scale (VAS). VAS is a simple and widely used tool for measuring subjective experiences such as pain. It typically consists of a 10 cm horizontal line, with the left end representing 'no pain' (0) and the right end representing 'worst imaginable pain' (10). The participant is asked to mark the point on the line that best reflects the intensity of their pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safe Practices When Positioning Patients in the Trendelenburg Position. AORN J. 2024 May;119(5):P9. doi: 10.1002/aorn.14134. No abstract available. PMID 38661435
- [Background] Celik B, Karayurt O, Ogce F. The Effect of Selected Risk Factors on Perioperative Pressure Injury Development. AORN J. 2019 Jul;110(1):29-38. doi: 10.1002/aorn.12725. PMID 31246295
- [Background] Engels D, Austin M, McNichol L, Fencl J, Gupta S, Kazi H. Pressure Ulcers: Factors Contributing to Their Development in the OR. AORN J. 2016 Mar;103(3):271-81. doi: 10.1016/j.aorn.2016.01.008. PMID 26924365
- [Background] Chen Y, Wang W, Qian Q, Wu B. Comparison of four risk assessment scales in predicting the risk of intraoperative acquired pressure injury in adult surgical patients: a prospective study. J Int Med Res. 2023 Oct;51(10):3000605231207530. doi: 10.1177/03000605231207530. PMID 37898108